CLINICAL TRIAL: NCT06863480
Title: THRIVE: Tocilizumab-aazg for Hemorrhage: Reduction of Ischemic Vascular Events
Brief Title: Tocilizumab-aazg for Hemorrhage: Reduction of Ischemic Vascular Events
Acronym: THRIVE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202201531
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Delayed Cerebral Ischemia
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- tocilizumab-aazg (TYENNE) (Experimental): Participants will receive tocilizumab-aazg 6mg/kg IV infusion drip on Day 0 following subarachnoid hemorrhage and enrollment in the trial.
  Interventions: Drug: tocilizumab-aazg (TYENNE)

INTERVENTIONS:
Drug: tocilizumab-aazg (TYENNE) — A single dose of tocilizumab-aazg (TYENNE) will be administered by intravenous drip.

SUMMARY:
In this study, tocilizumab-aazg (TYENNE) will be administered to see whether tocilizumab-aazg is safe in patients with a burst brain aneurysm and if it may prevent strokes in patients with a burst brain aneurysm.

DETAILED DESCRIPTION:
This is a prospective single-arm, single-center, open-label Phase 1 trial of tocilizumab-aazg 6mg/kg IV infusion drip on Day 0 in patients with aneurysmal subarachnoid hemorrhage. The trial is designed to demonstrate safety and to detect a signal that tocilizumab-aazg prevents delayed cerebral ischemia in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥18 years) with Hunt Hess Grade 1-3, Fisher score 3 or 3 and 4, aneurysmal subarachnoid hemorrhage within 24 hours of symptom onset (ruptured aneurysm confirmed by CTA, MRA or DSA)
* Must have external ventricular drain or lumbar drain, or plan to place an external ventricular drain or lumbar drain.
* Female subjects of child-bearing potential must have negative pregnancy test
* Signed informed consent from subject or legally authorized representative
* Able and willing to comply with followup visits
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, as defined below:

Women must remain abstinent or use non-hormonal contraceptive methods with a failure rate of 1% per year during the treatment period and for 2 months after the final dose of TYENNE. Women must refrain from donating or storing eggs during the same time period. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. If required per local guidelines or regulations, locally recognized acceptable methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.

The following are examples of adequate non-hormonal contraceptive methods: bilateral tubal ligation; male sterilization; copper intrauterine devices; male or female condom with or without spermicide; and cap, diaphragm, or sponge with spermicide.

• For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 2 months after the dose of TYENNE to avoid exposing the embryo. Men must refrain from donating sperm during this same period.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of preventing drug exposure. If required per local guidelines or regulations, information about the reliability of abstinence will be described in the local Informed Consent Form.

Exclusion Criteria:

* Evidence for vasospasm or DCI prior to study enrollment
* Hemodynamically unstable pre-enrollment
* Severe or unstable concomitant condition or disease (e.g., known significant neurological deficit, cancer, hematologic or coronary disease), or chronic condition (e.g., liver disease, kidney disease, or psychiatric disorder), that may increase the risk associated with study participation, or may interfere with the interpretation of study results
* Subjects who have received an investigational product or participated in another interventional clinical study within 30 days prior to enrollment.
* Known hypersensitivity or severe allergic reaction to tocilizumab and/or other biologics agents (i.e. shock, anaphylactic reactions)
* Serious infection defined as pneumonia, sepsis/septic shock, and neutropenic fever prior to enrollment
* Any previous treatment with IL-6 inhibitory therapy (e.g. satralizumab), alemtuzumab, etc.
* Total body irradiation or bone marrow transplantation within 6 months prior to baseline.
* Any previous treatment with anti-CD20, anti-CD19, eculizumab, belimumab, interferon, natalizumab, glatiramer acetate, fingolimod, teriflunomide or dimethyl fumarate within 6 months prior to baseline.
* Any previous treatment with anti-CD4, cladribine or mitoxantrone within 2 years prior to baseline
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 2 months after TYENNE administration
* Women of childbearing potential must have a negative serum pregnancy test result prior to initiation of study drug.
* Any surgical procedure (except for minor surgeries) within 4 weeks prior to baseline.
* Evidence of serious uncontrolled concomitant diseases that may preclude patient participation, such as: other nervous system disease, cardiovascular disease, hematologic/hematopoiesis disease, respiratory disease, muscular disease, endocrine disease, renal/urologic disease, digestive system disease, congenital or acquired severe immunodeficiency.
* Known active infection (excluding fungal infections of nail beds or caries dentium) within 4 weeks prior to baseline.
* History of diverticulitis that, in the principal investigator's opinion, may lead to increased risk of complications such as lower gastrointestinal perforation.
* Evidence of active or untreated latent tuberculosis (TB; excluding patients receiving chemoprophylaxis for latent TB infection).
* Evidence of active interstitial lung disease
* Receipt of any live or live attenuated vaccine within 6 weeks prior to baseline and throughout the duration of the study.
* History of malignancy within the last 5 years, including solid tumors, hematologic malignancies and in situ carcinoma (except basal cell and squamous cell carcinomas of the skin, or in situ carcinoma of the cervix uteri that have been completely excised and cured).
* Laboratory exclusion criteria (at screening):
* White blood cells (WBC) <3.0 x103/μL
* Absolute neutrophil count (ANC) <2.0 x103/μL
* Absolute lymphocyte count <0.5 x103/μL
* Platelet count <100 x 103/μL
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the upper limit of normal (ULN).
* Patient with known medical history at screening listed for the following must be excluded from this trial:
* Evidence of chronic active hepatitis B (HBV)
* Evidence of chronic active hepatitis C (HCV)
* Positive for hepatitis C virus (HCV) antigen
* Positive for hepatitis B surface antigen (HBsAg)
* Known HIV infection.
* Illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Poor peripheral venous access
* Serious infection requiring oral or IV antibiotics prior to screening
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* History or presence of an abnormal ECG that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third-degree atrioventricular heart block, or evidence of prior myocardial infarction

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with elevation of liver transaminases | up to 21 days
  Elevation of liver transaminase (ALT, AST) is defined as >5x upper limit of normal.
Number of participants with neutropenia | up to 21 days
  Neutropenia is defined as neutrophil count below 1 x 10^9/L.
Number of participants with decreased platelet count | up to 21 days
  Decreased platelet count is defined as a platelet count below the lower institutional limit of normal.
Frequency of observed and reported adverse events | baseline up to 90 days following the last administration of study treatment or study discontinuation/termination, whichever is earlier
  An adverse event will be defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational medicinal product (IMP) or other protocol-imposed intervention, regardless of attribution.
Frequency of death | baseline up to 90 days following the last administration of study treatment or study discontinuation/termination, whichever is earlier
  All deaths that occur during the protocol-specified AE reporting period, regardless of attribution, will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hoh, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health (UF Health), Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided